CLINICAL TRIAL: NCT04395092
Title: Haplo-identical Natural Killer (NK) Cells to Prevent Post-Transplant Relapse in AML and MDS (NK-REALM)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The sponsor decided to withdraw this study
Sponsor: Kiadis Pharma (Industry)
Collaborators: Blood and Marrow Transplant Clinical Trials Network (Network); National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BMT CTN 1803; U24HL138660 (NIH)
Record Dates: First submitted 2020-05-06; First posted 2020-05-20 (Actual); Last update posted 2021-06-22 (Actual); Status verified 2021-06

CONDITIONS: Acute Myeloid Leukemia (AML); Myelodysplastic Syndromes (MDS)
Keywords: K-NK002; NK cell therapy; AML; MDS
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — Transplantation Conditioning

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- K-NK002 (Experimental)
  Interventions: Biological: K-NK002; Procedure: Conditioning Regimen; Procedure: HaploBMT

INTERVENTIONS:
Biological: K-NK002 — K-NK002 will be administered intravenous (IV) on Day -2, Day +7 and Day +28.
  Part One (Safety run-in):
  An initial safety run-in to confirm the starting dose, and safety and tolerability of K-NK002;
  * Dose cohort 1 will include 3 patients who will receive a dose of K-NK002 at 1 x 10E7 NK cells per kg.
  * Dose cohort 2 will include 3 patients who will receive K-NK002 at 1 x 10E8 NK cells per kg.
  Part Two (Open Enrollment):
  Enrollment into the second part of the study (Open Enrollment) can begin following Part One, confirmation of dose and safety.
Procedure: Conditioning Regimen — From Day -7 to Day -3:
  * Melphalan: 140 mg/m2 (100mg/m2 in patients ≥ 60) on Day -7.
  * Fludarabine: 40 mg/m2 daily for 4 doses starting on days -7.
  * TBI: 2 Gy on Day -3.
Procedure: HaploBMT — Bone marrow is the only allowed graft source for patients enrolled in this clinical trial

SUMMARY:
This study is a Phase II, single arm, open label multicenter trial designed to investigate the use of haploidentical donor derived NK cells (K-NK002) for the treatment of patients with high-risk acute myeloid leukemia (AML) or myelodysplastic syndrome (MDS) who are undergoing haploidentical donor bone marrow transplantation (HaploBMT). K-NK002 is a NK cell product derived from peripheral blood leukocytes collected from a related donor (HLA-haploidentical matched) and enriched for NK cells with depletion of CD3+ T-lymphocytes (T-cells) followed by enriched ex-vivo expansion and administered to the patient prior to and following BMT.

DETAILED DESCRIPTION:
The study is a Phase II, single arm, open label, multicenter trial evaluating the cumulative incidence of relapse when K-NK002 is used for relapse mitigation in patients with high-risk AML and MDS receiving an allogeneic haploidentical bone marrow graft.

Part One (Safety run-in):

An initial safety run-in to confirm the starting dose, and safety and tolerability of K-NK002;

* Dose cohort 1 will include 3 patients who will receive a dose of K-NK002 at 1 x 10E7 NK cells per kg.
* Dose cohort 2 will include 3 patients who will receive K-NK002 at 1 x 10E8 NK cells per kg.

Part Two (Open Enrollment):

Enrollment into the second part of the study (Open Enrollment) can begin following Part One, confirmation of dose and safety.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 65 years.
2. Weight at least 45 kg.
3. Patients with AML must have high risk for disease relapse AND be in complete remission (CR), complete remission with incomplete hematologic recovery (CRi) or morphologic leukemia free state (MLFS). Patients with FLT3 internal tandem duplication (FLT3/ITD) mutation are eligible but must be made aware of alternative treatments available, e.g. tyrosine kinase inhibitor therapy as maintenance following transplantation.

   * AML patients must be in CR, CRi or a MLFS, as defined by ELN 2017.
4. Patients with high-risk MDS must meet one of the following criteria:

   * i. De novo MDS with intermediate/high/very high Revised International Prognostic Scoring System (R-IPSS) risk scores with

     1. Bone marrow blasts < 10%, AND
     2. Patients may be treatment-naïve, or have received prior treatment with hypomethylating agents or other therapies.
   * ii. Secondary/therapy-related MDS with bone marrow blasts < 10%.
5. Hematopoietic Cell Transplantation Comorbidity Index (HCT-CI) of 3 or less. The presence of prior malignancy will not be used to calculated HCT-CI for this trial to allow for the inclusion of patients with secondary or therapy-related AML or MDS.
6. Cardiac function: LVEF ≥ 45%.
7. Pulmonary function: DLCO corrected for hemoglobin ≥ 60% and FEV1 ≥ to 60% the predicted value.
8. Serum creatinine < 1.5 mg/dL or creatinine clearance by Cockroft-Gault ≥ to 50 ml/min
9. Hepatic ALT/AST < 5 x the institutional upper limit of normal (ULN) and total bilirubin < 1.5 mg/dl with conjugated (direct) bilirubin < 2 x ULN.

   a. Indirect hyperbilirubinemia due to Gilbert's syndrome is allowed including total bilirubin ≥ to 1.5 mg/dl
10. Karnofsky Performance Score ≥ to 70%.
11. Available first-degree related mismatched bone marrow donor [biologic parent, siblings (full or half) or children] as follows:

    1. Donor must be at least a full haplotype match (3/6 or 4/6 match only; 5/6 matches are not allowed) for human leukocyte antigen (HLA)-A and -B at intermediate (or higher) resolution, and -DRB1 at high resolution using DNA-based typing, AND
    2. Donor must be willing to donate bone marrow, AND
    3. Donor should be a candidate for bone marrow harvest, according to institutional standards.
12. Female patients must either:

    1. Be of non-childbearing potential, either postmenopausal or surgically sterilized.
    2. Or, if of childbearing potential agree to practice two effective methods of contraception or agree to completely abstain for intercourse from the time of signing the informed consent form through receiving immunosuppressive therapy post-transplant.
13. Male patients (even if surgically sterilized), and their female partners of childbearing potential must agree to use a highly effective contraception method.
14. Voluntary written consent obtained prior to the performance of any study-related procedure.

Exclusion Criteria:

1. Prior allogeneic transplant.
2. AML beyond CR2.
3. Patients who have a suitable HLA-matched related donor.
4. Donor specific anti-HLA antibodies (DSA) greater than 1000 MFI.
5. Hepatitis B, Hepatitis C, or HIV positive by PCR.
6. Liver cirrhosis or portal hypertension (successfully treated for Hepatitis B or C are recommended to be evaluated by elastography or liver biopsy to evaluated for cirrhosis).
7. Uncontrolled bacterial, viral or fungal infections (currently taking medication and with progression or no clinical improvement) at time of enrollment.
8. Another cancer in remission less than 2 yrs are not eligible. A history of a previously treated solid tumor whose remission status is 2 yrs or greater and are not receiving tumor directed therapy will be considered eligible. Hormonal therapy as a part of long-term maintenance post-malignancy is allowed.
9. Concurrent participation in another investigational clinical trial(s) with interventions which could influence relapse, GVHD, or viral reactivation.
10. Systemic corticosteroid use at the time of screening. Treatment with hydrocortisone for prevention of transfusion reactions are eligible, but use of methylprednisolone is not allowed.
11. Woman who are pregnant or lactating.
12. Any serious medical or psychiatric illness likely to interfere with participation in this clinical study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-11-13 (Actual); Primary Completion 2022-11 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Cumulative incidence of relapse | 1 year
  Cumulative incidence of relapse at 1 year

SECONDARY OUTCOMES:
Determine the safety and tolerability of K-NK002 through incidence of (Serious) Adverse Events. | 1-year post-transplant.
  As assessed by CTCAE v5.0, incidence of AEs and serious adverse events (SAEs) will be collected from the 1st dose of K-NK002 through 30 days after the last dose. In addition, any SAEs assessed as related to the investigational product that occurs after the 30-day follow-up period will be recorded till end of study.
Overall survival (OS). | 1-year post-transplant.
Rate of Non-Relapse Mortality (NRM). | 1-year post-transplant.
Relapse-free survival. | 1-year post-transplant.
GVHD-free survival. | 1-year post-transplant.
Cumulative incidence of grade II-IV and III-IV acute GVHD. | Day 100 post-transplant.
Cumulative incidence of chronic GVHD. | 1-year post-transplant.
Hematologic recovery as assessed according to neutrophil and platelet counts. | Up to day 100 post-transplant.
  * Neutrophil recovery: absolute neutrophil count (ANC) ≥ 500/mm3 for three consecutive measurements on three different days.
  * Platelet recovery: the first day of a sustained platelet count ≥ 20,000/mm3 or ≥50,000/mm3 with no platelet transfusions in the preceding seven days.
Donor cell engraftment. | Days 28 and 100 post-transplant.
  Frequencies and percentage of patients with full (>95%), mixed (5-95%), or low (<5%) chimerism at each time point. Mixed and full chimerism will be evidence of donor cell engraftment.
Primary and secondary graft failure as measured by neutrophil count. | By days 28 and 100 post-transplant.
Overall toxicity. | From 1st dose of K-NK002 to 30 days after last dose.
  Incidence of all grade 1-5 AE from 1st dose of K-NK002 to 30 days after the last dose of K-NK002 according to CTCAE v5.0.
Cumulative incidence of CMV reactivation and symptomatic BKV hemorrhagic. cystitis. | Days 100 and 180 post-transplant.

CONTACTS AND LOCATIONS:
Overall Officials: Sumithira Vasu, MD, Study Chair — Ohio State University; Richard Champlin, MD, Study Chair — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - Northside Hospital, Atlanta, Georgia
  - MD Anderson, Houston, Texas

IPD SHARING:
Plan to Share IPD: No